CLINICAL TRIAL: NCT03699176
Title: A Randomized, Parallel-group, Double-blind Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of Vilaprisan in Subjects With Uterine Fibroids
Brief Title: Assessment of Safety and Efficacy of Vilaprisan in Subjects With Uterine Fibroids
Acronym: ASTEROID 7
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No patient was recruited, study withdrawn for feasibility reasons.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19434
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — vilaprisan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vilaprisan (Experimental): 2 treatment periods of 12 weeks without a break
  Interventions: Drug: Vilaprisan (BAY1002670)
- Placebo (Placebo Comparator): 2 treatment periods of 12 weeks without a break
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — 2 mg, once daily, oral
  Arms: Vilaprisan
Drug: Placebo — Once daily, oral
  Arms: Placebo

SUMMARY:
The primary objective of this study is to show superiority of vilaprisan in the treatment of heavy menstrual bleeding (HMB) in subjects with uterine fibroids compared to placebo.The secondary objectives of this study are to additionally evaluate the efficacy and safety of vilaprisan in subjects with uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 years or older at the time of Visit 1
* Diagnosis of uterine fibroid(s) documented by ultrasound at screening with at least 1 fibroid with largest diameter of ≥ 30 mm (alternatively, of 30 mm or more)
* Heavy menstrual bleeding (HMB) in at least 2 bleeding periods during the screening period each with blood loss volume of >80.00 mL documented by the menstrual pictogram (MP)
* Use of an acceptable non-hormonal method of contraception
* An endometrial biopsy performed during the screening period, without significant histological disorder such as endometrial hyperplasia (including simple hyperplasia) or other significant endometrial pathology

Exclusion Criteria:

* Pregnancy or lactation (less than 3 months since delivery, abortion, or lactation before start of treatment)
* Hypersensitivity to any ingredient of the study drugs
* Hemoglobin values ≤6 g/dL or any condition requiring immediate blood transfusion (subjects with hemoglobin values ≤10.9 g/dL will be recommended to use iron supplementation)
* Any diseases, conditions, or medications that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug including
* Abuse of alcohol, drugs, or medicines (eg: laxatives)
* Undiagnosed abnormal genital bleeding
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Amenorrhea (yes/no) | Up to 24 weeks (The last 28 days of treatment period 2)
  Defined as menstrual blood loss (MBL) <2 mL (based on menstrual pictogram)

SECONDARY OUTCOMES:
Heavy menstrual bleeding (HMB) response (yes/no) | Up to 24 weeks (the last 28 days of treatment period 2)
  Defined as blood loss <80.00 mL during the last 28 days of treatment and >50% reduction compared to baseline
Time to onset of amenorrhea | Up to 24 weeks
  Onset of amenorrhea is defined by the first day for which the menstrual blood loss for all subsequent 28-day periods up to the end of the treatment period is <2mL.
Time to onset of controlled bleeding | Up to 24 weeks
  Onset of controlled bleeding is defined by the first day for which the menstrual blood loss for all subsequent 28-day periods up to the end of the treatment period is <80.00 mL.
Absence of bleeding (spotting allowed) based on the Uterine Fibroid Daily Bleeding Diary (UF-DBD) | Up to 24 weeks (the last 28 days of treatment period 2)
Endometrial histology (eg, benign endometrium, presence or absence of hyperplasia or malignancy) | Up to 36 weeks
Endometrial thickness | Up to 36 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Funabashi Municipal Medical Center, Funabashi, Chiba
  - Matsudo City General Hospital, Matsudo, Chiba
  - Ena Odori Clinic, Sapporo, Hokkaido
  - Tokeidai Memorial Clinic, Sapporo, Hokkaido
  - Asahi clinic, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Unoki Clinic, Kagoshima
  - Japanese Red Cross Kumamoto Hospital, Kumamoto